CLINICAL TRIAL: NCT03712774
Title: Prospective Observational Trial to Evaluate Quality of Life After Neoadjuvant or Definitive Chemoradiation in Patients With Esophageal Cancer
Acronym: ESOCARE
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Falk Roeder, Consultant, Ludwig-Maximilians - University of Munich
Other Study IDs: V1 08_2018
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Quality of Life; Chemoradiation; Esophageal Cancer
Keywords: quality of life; neoadjuvant; definitive; chemoradiation; esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoadjuvant chemoradiation: Patient with esophageal Cancer treated by neoadjuvant chemoradiation followed by surgery will be longitudinally evaluated by questionaires EORTC QLQ C30, EORTC QLQ OES-18 and EORTC OG-25
  Interventions: Other: EORTC QLQ C30; Other: EORTC QLQ OES-18; Other: EORTC OG-25
- definitive chemoradiation: Patient with esophageal Cancer treated by definitive chemoradiation will be longitudinally evaluated by questionaires EORTC QLQ C30, EORTC QLQ OES-18 and EORTC OG-25
  Interventions: Other: EORTC QLQ C30; Other: EORTC QLQ OES-18; Other: EORTC OG-25

INTERVENTIONS:
Other: EORTC QLQ C30 — standardized questionaire
Other: EORTC QLQ OES-18 — standardized questionaire
Other: EORTC OG-25 — standardized questionaire

SUMMARY:
Prospective observational study to evaluate the Quality of life based on standardized EORTC questionaires as well as toxicities, functional and oncological outcomes in patients treated with neoadjuvant or definitive chemoradiation for esophageal Cancer.

DETAILED DESCRIPTION:
Prospective observational study to evaluate the Quality of life based in patients treated with neoadjuvant or definitive chemoradiation for esophageal Cancer. QoL will be evaluated by standardized EORTC questionaires. Acute and late toxicity will be assessed according to CTCAE 4.03. Outcome measures will include local Control, distant Control, freedom from Treatment failure and overall survival. Correlations are planned between Patient- and physician-assessed functional Outcome.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven esophageal Cancer (SCC or adenocarcinoma) without distant metastases (except supraclavicular nodes)
* indication for neoadjuvant or definitive chemoradiation using either cisplatin/5-FU or carboplatin/paclitaxel with curative intent
* age >= 18 years
* written informed consent
* ability to answer the standardized questionaires according to the treating physician

Exclusion Criteria:

* age < 18 years
* Treatment with palliative intent
* distant metastases (except supraclavicular nodes)
* second malignancy
* Prior systemic treatment for esophageal Cancer
* Treatment in an interventional study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: see eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | planning CT (day 0), week 4 of RT, 6 weeks after end of RT, 3 months after end of RT, 6 months after end of RT, 12 months after end of RT, 24, 36, 48, and 60 months after end of RT
  Quality of life measured by standardized EORTC questionaires

SECONDARY OUTCOMES:
Local control | 3 months after end of RT, 6 months after end of RT, 9 months after end of RT, 12 months after end of RT, 24,36,48,60 months after end of RT
  Absence of local progression
Distant Control | 3 months after end of RT, 6 months after end of RT, 9 months after end of RT, 12 months after end of RT, 24,36,48,60 months after end of RT
  Absence of distant metastases
freedom from treatment failure | 3 months after end of RT, 6 months after end of RT, 9 months after end of RT, 12 months after end of RT, 24,36,48,60 months after end of RT
  Absence of local and distant failure
Overall survival | 3 months after end of RT, 6 months after end of RT, 9 months after end of RT, 12 months after end of RT, 24,36,48,60 months after end of RT
  Absence of death by any cause
acute toxicity | end of RT, 6 weeks after end of RT, 3 months after end of RT
  acute toxicity scored according to CTCAE 4.03
late toxicity | 6 months after end of RT, 9 months after end of RT, 12, 24, 36, 48, 60 months after end of RT
  late toxicity scored according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Falk Roeder, MD, Principal Investigator — Ludwig-Maximilians Universität München
Locations (1):
- Department of Radiation Oncology, University Hospital, LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No